CLINICAL TRIAL: NCT04853628
Title: ALERTA ALCOHOL: The Development and Evaluation of an Animation- Versus Text-based Computer-tailored Game Intervention to Prevent Alcohol Consumption and Binge Drinking in Adolescents
Brief Title: An Animation- Versus Text-based Computer-tailored Game Intervention to Prevent Alcohol Consumption in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Delegación del Gobierno para el Plan Nacional sobre Drogas (Unknown); Maastricht University (Other)
Responsible Party: Principal Investigator, Marta Lima Serrano, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University of Seville (Spain)
Record Dates: First submitted 2021-04-09; First posted 2021-04-21 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Drinking; Binge Drinking; Adolescent Behavior
Keywords: Alcohol use; Binge drinking; High-intensity drinking; Adolescents; Web-based interventions; Computer-tailoring; Animation
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking; Adolescent Behavior | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: The study is performed in 24 high schools from Andalusia (southern Spain), which are randomized either to the experimental (EC-1, EC-2) or the control conditions (CC). The EC-1 receives Alerta Alcohol, with personalized health advice, using textual feedback and several gamification techniques; and consists of nine sessions (performing seven of them at the high school): session 1 or baseline, sessions 2 and 3 where adolescents are provided with answers related to their views to provide highly specific feedback regarding their knowledge, risk perception, self-esteem, attitude, social influence and self-efficacy; sessions 4, 5, 7 and 8 are reinforcement sessions (booster sessions) and sessions 6 and 9 are follow-up questionnaires at six and twelve months. The EC-2 receives Alerta Alcohol 2.0, using animated videos and new gamification strategies. The CC just completes the baseline and the evaluation questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alerta Alcohol (Experimental): The EC-1 receives Alerta Alcohol, which consists of session 1 or baseline, two sessions in three scenarios: at home, celebrations, and public places, and two follow-up evaluations. The adolescents are provided with answers related to their views of each scenario; this information is used to provide highly specific feedback regarding their knowledge, risk perception, self-esteem, attitude, social influence (modelling, norms and social pressure), self-efficacy and action plans. In addition, four booster sessions are given at home to reinforce the contents of the three scenarios. Evaluations take place after six and twelve months.
  Interventions: Behavioral: Alerta Alcohol
- Alerta Alcohol 2.0 (Experimental): The EC-2 receives an improved version of Alerta Alcohol (Alerta Alcohol 2.0) using animated videos and new gamification strategies. Evaluations take place after six and twelve months.
  Interventions: Behavioral: Alerta Alcohol 2.0
- Control condition (No Intervention): The CC just completes the baseline and the evaluation questionnaires and then they are allowed to receive the intervention as well (as a waiting list). Evaluations take place after six and twelve months from baseline.

INTERVENTIONS:
Behavioral: Alerta Alcohol — The intervention consists of preventive messages about the benefits of not consuming alcohol, reducing the positive attitudes and encouraging the negative attitudes towards alcohol drinking and BD, as well as social influence and self-efficacy, by personalized feedback. Skills and action plans are encouraged to help the student to reject BD. This information is presented through different tailored text messages. Moreover, several gamification strategies are used (i.e. offering a challenge, giving different stories and the use of avatars in these stories that take place in three different scenarios: at home, at celebrations and in public places).
  Other Names: A text-based computer-tailored game intervention
  Arms: Alerta Alcohol
Behavioral: Alerta Alcohol 2.0 — The intervention consists of preventive messages about the benefits of not consuming alcohol, reducing the positive attitudes and encouraging the negative attitudes towards alcohol drinking and BD, as well as social influence and self-efficacy, by personalized feedback. Skills and action plans are encouraged to help the student to reject BD. This information is presented through different animated videos. Moreover, new gamification strategies are added (i.e. giving rewards and allocating points that can be accumulated and shown in a progress ranking) to those already used in Alerta Alcohol.
  Other Names: An animation-based computer-tailored game intervention
  Arms: Alerta Alcohol 2.0

SUMMARY:
This study consists in the design, implementation and evaluation of an animation (Alerta Alcohol 2.0)- versus text-based (Alerta Alcohol) computer-tailored game intervention aimed to prevent alcohol consumption and binge drinking (BD) in Spanish adolescents. A Cluster Randomized Controlled Trial (CRCT) is conducted to test the effectiveness of Alerta Alcohol versus Alerta Alcohol 2.0 in students aged 14 to 19 years across 24 high schools from Andalusia (southern Spain), which are randomized either to the experimental (EC-1, EC-2) or the control conditions (CC).

DETAILED DESCRIPTION:
Alcohol use and misuse, and particularly, BD in adolescents are a highly prevalent healthcare problem that associates physical and mental health complications and community implications. The Alerta Alcohol and Alerta Alcohol 2.0 programs are based on the I-Change Model. A CRCT is carried out. The schools from Andalusia are randomized either to the experimental (EC-1, EC-2) or the control conditions (CC). The EC-1 receives an online intervention (Alerta Alcohol, which has adapted from a previous version) with personalized health advice, using textual feedback and several gamification techniques, and consists of nine sessions (performing seven of them at the high school): session 1 or baseline, sessions 2 and 3 where adolescents are provided with answers related to their views to provide highly specific feedback regarding their knowledge, risk perception, self-esteem, attitude, social influence and self-efficacy; sessions 4, 5, 7 and 8 are reinforcement sessions (booster sessions) and sessions 6 and 9 are follow-up questionnaires at six and twelve months. The EC-2 receives an improved version of Alerta Alcohol (Alerta Alcohol 2.0) using animated videos and new gamification strategies. The CC just completes the baseline and the evaluation questionnaires and then they are allowed to receive the intervention as well (as a waiting list). To test the effectiveness, the primary outcome is BD within 30 days prior to evaluation and alcohol use (high-intensity drinking, weekly and any consumption) in the previous week as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Students aged 14 to 19 years.
* Enrolled in Andalusian public or private high schools.
* Access to the Internet at the schools and the use of computer, mobile or tablet is allowed.
* Access to the Internet in their homes.

Exclusion Criteria:

* Language barriers.
* Previous participation in prevention programs for BD.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2625 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change on the prevalence of binge drinking | 6 months after the baseline
  Change on the prevalence of binge drinking (4/5 standard drink units or standard glasses of alcohol in one occasion for a girl/boy) within 30 days prior to evaluation.
Change on the prevalence of binge drinking | 12 months after the baseline
  Change on the prevalence of binge drinking (4/5 standard drink units or standard glasses of alcohol in one occasion for a girl/boy) within 30 days prior to evaluation.

SECONDARY OUTCOMES:
Change on the prevalence of high-intensity drinking | 6 months after the baseline
  Change on the prevalence of high-intensity drinking (8/10 standard drink units or standard glasses of alcohol in one occasion for a girl/boy) within the 7 days prior to evaluation.
Change on the prevalence of high-intensity drinking | 12 months after the baseline
  Change on the prevalence of high-intensity drinking (8/10 standard drink units or standard glasses of alcohol in one occasion for a girl/boy) within the 7 days prior to evaluation.
Change on the average of weekly consumption | 6 months after the baseline
  Change on the average of the total number of glasses consumed within the 7 days prior to evaluation.
Change on the average of weekly consumption | 12 months after the baseline
  Change on the average of the total number of glasses consumed within the 7 days prior to evaluation.
Change on the prevalence of any consumption | 6 months after the baseline
  Change on the prevalence of any consumption
Change on the prevalence of any consumption | 12 months after the baseline
  Change on the prevalence of any consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Marta Lima Serrano, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with other researchers through publications in scientific journals and conferences/congresses.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From 2021.
Access Criteria: The Access Criteria will be the one exposed by the scientific journals where the results of the study will be published.